CLINICAL TRIAL: NCT01247649
Title: Assessing Continuous Non- Invasive Blood Glucose Sensor- Physical Logic AG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: rmc006039ctil
Record Dates: First submitted 2010-11-21; First posted 2010-11-24 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Type 1 Diabetes
Keywords: Continuous glucose monitoring system; Non invasive; Type 1 diabetes; Dielectric spectroscopy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental): Patients will be monitored to assess continuous blood glucose levels using the study device (Physical Logic) and reference methods, during 2-3 clinic visits, lasting 6-8 hours each
  Interventions: Device: Physical Logic Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Physical Logic Continuous Glucose Monitoring System — Patients will be monitored to assess continuous blood glucose levels using the study device (Physical Logic) and reference methods, during 2-3 clinic visits, lasting 6-8 hours each

SUMMARY:
The present study is aimed to evaluate the feasibility of a new noninvasive method to measure continuous glucose values using electromagnetic radiation.

DETAILED DESCRIPTION:
The non invasive continuous glucose sensing system of Physical Logic is based on a vector network analyzer (VNA), which monitor blood glucose through propriety sensors.Dielectric spectroscopy is an analytical technique whereby the electromagnetic radiation is affected by the electric dipole moment of the sample it interacts with. This method utilizes the change in the impedance of the antenna to measure the change in the relaxation processes of the interrogated medium.

The VNA (vector network analyzer) , which emits non irradiating electromagnetic waves in very low power emission, is connected via standard coaxial cables to propriety sensors that are attached to the patient skin without direct contact.

Study objective:

To evaluate the feasibility of a new noninvasive method to measure continuous glucose values using electromagnetic radiation.The glucose values generated by the investigational non invasive devise will be compared to glucose reading of a reference devise, which measure blood glucose levels at the subcutaneous tissue.

During the study we will evaluate the reliability of the study device under the conditions of alter blood glucose values in the range of 50-400 mg/dl:

ELIGIBILITY:
Inclusion Criteria:

1. Signing an inform consent form
2. Type 1 diabetes diagnosed at least 12 months prior to study inclusion
3. Age > 18 years old
4. Willing to perform all study related procedures

Exclusion Criteria:

1. Known or suspected allergy to the sensor or one of its components
2. Psychiatric disorder
3. Patients with one or more of the following diseases: malignancy, myocardial insufficiency, nephrologic disease or any other chronic disease
4. Patients who are not willing or are not capable of performing the protocol requirements
5. Participating in another study that includes investigational drug or investigational equipment
6. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Correlation between continuous glucose measurements using study device and YSI(yellow springs instrument) | up to 24 weeks
  Correlation between continuous glucose measurements using study device (Physical Logic) and YSI(yellow springs instrument)at variable glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Revital Nimri, Dr, Principal Investigator — Schenider Children's Medical
Locations (1):
- Schneider Children's Medical center, Petah Tikva, Israel